CLINICAL TRIAL: NCT00257049
Title: A Multicenter, Active-Controlled, Randomized Study To Evaluate The Safety And Efficacy Of Levofloxacin Versus Ceftriaxone Sodium Or Cefuroxime Axetil In The Treatment Of Community-Acquired Pneumonia In Adults
Brief Title: A Study of the Safety and Effectiveness of Levofloxacin Compared With Ceftriaxone Sodium or Cefuroxime Axetil in the Treatment of Adults With Pneumonia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005491
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-11

CONDITIONS: Pneumonia
Keywords: Pneumonia; lung inflammation; bacterial pneumonia; lung diseases; respiratory tract infections; antibacterial agents; quinolones; levofloxacin
MeSH Terms: conditions — Pneumonia; Pneumonia, Bacterial; Lung Diseases; Respiratory Tract Infections | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is evaluation of the safety and effectiveness of levofloxacin, an antibiotic, compared with ceftriaxone sodium or cefuroxime axetil in the treatment of adults with pneumonia.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel group, multicenter study to determine the safety and effectiveness of levofloxacin (488 mg once daily by mouth or 500 mg administered intravenously once daily for 7 - 14 days) compared with ceftriaxone sodium (1 - 2 grams administered into a vein or muscle once daily or in divided doses twice daily for 7 - 14 days) or cefuroxime axetil (500 mg by mouth twice daily for 7 - 14 days) in adults with community-acquired pneumonia. The study consists of 4 visits: one visit for screening and enrollment, and 3 visits for assessment of safety and effectiveness (one visit on Day 2 - 4 [on-therapy], one visit [post-therapy] 5 - 7 days after the last dose of the study drug, and one visit [post-study] 21 - 28 days after the last dose of the study drug). The total duration of patient participation in the study is approximately 6 weeks. Levofloxacin is an antibacterial agent used for the treatment of many types of infections in adults. The purpose of this study is to compare the safety and effectiveness of levofloxacin with other frequently used antibiotics (ceftriaxone sodium or cefuroxime axetil) in the treatment of adults with pneumonia acquired in the community. The primary efficacy assessment is the clinical response 5 - 7 days after the last dose of study drug, (categorized as cured, improved, or failed) based upon changes in signs and symptoms, and changes in x-ray findings, Safety evaluations (incidence of adverse events, physical examination, and laboratory tests) are performed throughout the study. Cost-effectiveness is also assessed for the study drugs. The study hypothesis is that treatment with levofloxacin will be at least as effective as ceftriaxone sodium or cefuroxime axetil in treating patients with pneumonia acquired in the community, and that it will be well tolerated. Levofloxacin 488 mg by mouth once daily or 500 mg intravenously once daily; ceftriaxone sodium (1 - 2 grams administered into a vein or muscle once daily or in divided doses twice daily); or cefuroxime axetil (500 mg by mouth twice daily). Treatment duration is 7 - 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pneumonia based upon clinical signs and symptoms of a lower respiratory tract infection including at least 2 of the following: fever, cough, greenish-yellow mucus produced on coughing, chest pain, shortness of breath, or evidence of decreased lung function during the physical examination
* has chest x-ray findings consistent with acute pneumonia
* previously received antibiotics for pneumonia if the duration of therapy was <= 24 hours, or if greater than 24 hours, but without improvement or stabilization with that therapy.

Exclusion Criteria:

* Previous allergic or serious adverse reaction to any antibiotic similar to those used in this study or to penicillin
* collection of pus in the cavity between the lung and the membrane that surrounds it
* has cystic fibrosis
* has a lung infection due to fungus, bacteria, or virus known prior to the start of the study to be resistant to any of the study drugs
* has severe kidney failure, decrease in white blood cell count, seizure disorder, or an unstable psychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Actual)
Dates: Start 1984-01; Study Completion 1995-01 (Actual)

PRIMARY OUTCOMES:
Clinical response rate (reduction in signs and symptoms, improvement in x-ray findings) at post-therapy (5 - 7 days after the last dose of study drug).

SECONDARY OUTCOMES:
Rate of elimination of disease-causing bacteria, by patient, and by type of bacteria; incidence of adverse events; changes in physical examination and laboratory tests after treatment with study drug

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety and effectiveness of levofloxacin compared with ceftriaxone sodium or cefuroxime axetil in the treatment of adults with pneumonia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=656&filename=CR005491_CSR.pdf